CLINICAL TRIAL: NCT06290505
Title: PALEO: Phase II Clinical Trial of Chemoradioimmunotherapy for the ALleviation of oEsOphageal Cancer Complications
Brief Title: A Trial of Palliative Chemotherapy, Radiation and Immune Treatment for Oesophageal Cancer: PALEO Study
Acronym: PALEO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALEO
Record Dates: First submitted 2023-10-18; First posted 2024-03-04 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will receive 2 weeks of therapy with concurrent hypofractionated radiotherapy (30Gy/10#), weekly carboplatin (AUC2), weekly paclitaxel (50mg/m2) and durvalumab (1500mg) intravenously every 4 weeks, followed by durvalumab monotherapy continuing at 1500mg intravenously every 4 weeks until disease progression or 24 months of therapy. One to five metastases will be treated with stereotactic radiotherapy (24Gy/3#) 4 weeks after the completion of the chemoradiotherapy to the primary tumour. Monitoring of adherence to treatment will be done by attendance at booked appointments
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab will be supplied by AstraZeneca as a 500 mg vial concentrate for solution for infusion. The solution contains 50 mg/mL durvalumab, 26 mM histidine/histidine-hydrochloride, 275 mM trehalose dihydrate, and 0.02% weight/volume (w/v) polysorbate 80; it has a pH of 6.0 and density of 1.054 g/mL. The label-claim volume is 10 mL.
  Durvalumab is a sterile, clear to opalescent, colorless to slightly yellow solution, free from visible particles.
  Investigational product vials are stored at 2°C to 8°C and must not be frozen. Investigational product must be kept in original packaging until use to prevent prolonged light exposure.
  Other Names: Imfinzi

SUMMARY:
The purpose of this study is to investigate the effects of the addition of the stereotactic body radiotherapy and durvalumab to a well tolerated 2 week chemotherapy and radiation treatment regimen in people with esophageal cancer that is locally advanced or has spread to another area of the body (metastasized).

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of the addition of the stereotactic body radiotherapy and durvalumab to a well tolerated 2 week chemotherapy and radiation treatment regimen in people with esophageal cancer that is locally advanced or has spread to another area of the body (metastasized).

Who is it for?

Participant may be eligible for this study if participant is an adult who has cancer of the esophagus or gastro-esophageal junction that is locally advanced or has spread to other parts of the participant's body.

Study details

All participants in this study will receive 10 treatments of radiotherapy to the primary esophageal cancer, with one treatment given on each working day for two weeks. In addition, all participants will receive chemotherapy (including carboplatin and paclitaxel) given intravenously once per week for the same two weeks as the radiotherapy. Durvalumab, an immune therapy, received intravenously; will be given every four weeks from the beginning of radiation therapy.

After this participants will continue to receive immune therapy (durvalumab), received intravenously once every 4 weeks for up to 24 months or until the cancer worsens. If participants have a metastatic tumour, they will also be given 3 doses of radiotherapy in one week. This radiotherapy will be received 4 weeks after the initial radiotherapy is completed.

Safety blood tests will be collected throughout the study (every two weeks from week 2 of treatment and then every four weeks from week 9 throughout the treatment and at other times if clinically indicated). CT scans to evaluate the response to treatment will be done every 6 weeks up to week 24 of treatment and then every 12 weeks or until the cancer worsens. Study participants will also be asked to complete some questionnaires about their wellbeing and nutritional status periodically throughout the study.

It is hoped that this trial can help determine if this chemotherapy with immune therapy and radiotherapy combination is effective in increasing the ability of the body's immune system to prevent worsening of the cancer and improve swallowing.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females > 18 years of age.
2. Biopsy proven adenocarcinoma or squamous cell carcinoma of the esophagus or gastro-oesophageal junction
3. Oligometastatic disease (1-5 lesions outside the primary tumour radiotherapy field on FDG-PET scan), or locoregionally advanced disease unsuitable for either surgical resection or radical chemoradiotherapy
4. Symptomatic dysphagia (Mellow score greater than 0)
5. ECOG performance status 0-2
6. Anticipated life expectancy of greater than 12 weeks.
7. Body weight of greater than 30kg.
8. Adequate bone marrow function, with values within the ranges specified below. Blood transfusions are permissible.

   1. White blood cell count greater than or equal to 2 x (10 to the power of 9)/L
   2. Absolute neutrophil count greater than or equal to 1.5 x (10 to the power of 9)/L
   3. Platelets greater than or equal to 100 x (10 to the power of 9)/L
   4. Haemoglobin greater than or equal to 90g/L
9. Adequate liver function, with values within the ranges specified below:

   1. Alanine transferase less than or equal to 2.5 x upper limit of normal (ULN)
   2. Aspartate transferase less than or equal to 2.5 x ULN
   3. Total bilirubin less than or equal to 1.5 x ULN (except patients with Gilbert's Syndrome, who can have total bilirubin less than or equal to 5 x ULN)
10. Adequate renal function, with values within the ranges specified below. Note that an estimated renal function of greater than 125mL/min by the Cockroft-Gault formula must not be used for carboplatin dosing, and must instead be determined using a direct method.

    1. Serum creatinine less than or equal to 1.5 x ULN
    2. Creatinine clearance (CrCl) greater than or equal to 40 mL/min using Cockroft-Gault formula
11. Tumour tissue (formalin-fixed, paraffin embedded) should be available for PD-L1 and mismatch repair (MMR) protein expression and can be provided as a block or slides (archival tissue is acceptable). Blocks prepared from cytological samples, where tumour cell number is sufficient, are also acceptable. Patients will not be selected by PD-L1 or MMR status.
12. Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments.
13. Signed, written and informed consent.

Exclusion Criteria:

1. Bulky or organ-threatening metastatic disease requiring upfront higher dose chemotherapy in the judgement of the treating clinician.
2. Known tumour HER2 positivity (IHC 2+ or more and HER2 gene amplification on in situ hybridisation) if oligometastatic disease.
3. Previous systemic therapy for oesophageal or GOJ carcinoma.
4. Previous thoracic radiotherapy. Prior palliative radiotherapy to bony metastases is permitted.
5. Esophageal stent in situ.
6. Known tracheo-oesophageal fistula.
7. Known leptomeningeal or brain metastases.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to first day of study treatment. Note: Local surgery of isolated lesions for palliative intent is permitted.
9. History of another malignancy within the last 3 years, with the exception of adequately treated non-melanomatous skin cancer, carcinoma in situ and superficial transitional cell carcinoma of the bladder.
10. Prior therapy with an anti-PD1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways.
11. Sensory neuropathy of grade 2 or higher severity per CTCAE v5.0.
12. History of allergy or hypersensitivity to study drug components, or other contraindications to any of the study drugs. Active or prior documented autoimmune disorders (including inflammatory bowel disease [e.g., ulcerative colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc). Patients with the following conditions are exceptions to this criterion:

    1. Vitiligo or alopecia.
    2. Hypothyroidism (e.g., following Hashimoto syndrome) stable on thyroid hormone replacement.
    3. Any chronic skin condition (e.g. psoriasis) that does not require systemic therapy.
    4. Type 1 diabetes mellitus.
    5. Coeliac disease controlled by diet alone.

    Patients without active autoimmune disease in the last 5 years may also be included but only after consultation with the Chief Principal Investigators.
13. Any condition requiring continuous systemic treatment with either regular corticosteroids (>10mg daily prednisone or equivalent dose of an alternative corticosteroid) or other immunosuppressive medications within 14 days of study drug administration. Intranasal, inhaled or topical steroids, and adrenal replacement steroid doses >10mg daily oral prednisone equivalent, are permitted in the absence of active autoimmune disease.
14. Positive test for hepatitis B surface antigen (HBsAg) indicating acute or chronic infection. Participants with a past or resolved HBV infection (defined as the presence of anti-HBc and absence of HBsAg) are eligible.
15. Positive test for hepatitis C virus antibody (HCV antibody) , unless polymerase chain reaction is negative for HCV RNA.
16. History of other significant, or active, infection, including HIV or tuberculosis (TB). HIV testing is not mandatory unless clinically indicated. Clinical evaluation for active TB may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice.
17. Receipt of a transplanted solid organ (kidney, liver, heart or lung) or of an allogeneic bone marrow transplant.
18. Receipt of a live attenuated vaccine within 30 days prior to registration.
19. Use of alternative or traditional medicines within 14 days prior to registration.
20. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events or compromise the ability of the patient to give written informed consent.
21. Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal, infertile, or use a reliable means of contraception to avoid pregnancy for 90 days after the last dose of durvalumab. Women of childbearing potential must have a negative pregnancy test within 24 hours prior to trial registration. Men must have been surgically sterilized or use a double barrier method of contraception if they are sexually active with a woman of childbearing potential for a period of 180 days after the last dose of durvalumab and chemotherapy, or 90 days after the last dose of durvalumab monotherapy (whichever is the longer time period). Sperm donation is not permitted for 180 days after the last dose of durvalumab and chemotherapy, or 90 days after the last dose of durvalumab monotherapy (whichever is the longer time period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate is the proportion of patients alive and progression free (the cancer has not worsened) assessed by CT scan and clinical review. | 6 months
  The interval from the date of participant registration to the date of a progression free survival event:
  1. date of the first CT scan to show disease progression
  2. patient is judged to have progressed by the responsible investigator (in the event that no RECIST assessment is available)
  3. death occurs.

SECONDARY OUTCOMES:
Duration of dysphagia relief | Mellow score will be assessed at days 1, 8, 15, 29, 43, 57 and then every 4 weeks thereafter until the end of treatment visits (30days after the last dose).
  Maintenance of Mellow score at least 1 point above baseline. Mellow score may be optionally assessed at days 22, 36 and 50 if the participants attend the clinic for any other unscheduled visit. Mellow score ranges from grade 0-4. Grade 0 indicating no dysphagia and grade 4 indicating inability to swallow.
Nutritional status | To be administered by a qualified dietician from date of randomisation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 weeks.
  Determined by clinical review and collected from the participant using the scored Patient-generated subjective global assessment (PG_SGA) tool.
Quality of life change using the - European organisation for the research and treatment of cancer quality of life questionnaire QLQ-C30 | Through study completion, an average of 1 year, using the 4-point ordinal scale - not at all, a little, quite a bit and very much
  Assessment of European organisation for the research and treatment of cancer quality of life questionnaire QLQ-C30
Quality of life change using the - European organisation for the research and treatment of cancer quality of life questionnaire QLQ-OES18 | Through study completion, an average of 1 year, using the 4-point ordinal scale - not at all, a little, quite a bit and very much
  Assessment of European organisation for the research and treatment of cancer quality of life questionnaire QLQ-OES18
Response rate in metastatic lesions | Assessment with imaging scans is performed at baseline then every 6 weeks while in treatment, then every 12 weeks until disease progression or date of death from any cause, whichever came first, assessed up to 96 weeks.
  Assessed using radiological imaging with Contrast CT Scan (chest and abdomen, + neck)
Physician graded toxicity | Assessed from baseline to 90 days following last treatment dose.
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
SAE Rate | Days 1, 8, 15, 29, 43, 57 and then every 4 weeks thereafter until to 100 days after last dose durvalumab regardless of relationship to drug.
  Assessed as reported by the participant and by clinician assessment from consent signing to 100 days after last dose of durvalumab regardless of relationship to drug. Adverse events will be documented in the patient medical record. A serious adverse event (SAE) is any untoward medical occurrence that at any dose: 1) results in death, 2) is life-threatening (i.e. the participant is at risk of death at the time of the event), 3) requires inpatient hospitalisation or prolongation of existing hospitalisation, 4) results in persistent or significant disability or incapacity, 5) is a congenital anomaly/birth defect, 6) other important medical events which may jeopardize the patient or may require intervention to prevent one of the listed outcomes in the definition above, which, in the opinion of the Investigator, are likely to become serious if untreated.
Overall survival. | Throughout study completion, average 2 years
  Overall survival will be reported with Kaplan Meier curves and summarized by their medians, and proportions event-free

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Day, Dr, Study Chair — Calvary Mater Newcastle; Jared Martin, Professor, Study Chair — Calvary Mater Newcastle
Locations (9):
- Australia (8):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Border Medical Oncology, Albury, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - St Vincent's Hospital, Fitzroy, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Auckland Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
Data sharing is encouraged and will be considered following submission of a concept for a secondary analysis